CLINICAL TRIAL: NCT00318123
Title: Multicentre, Open Label, Prospective, Randomised Clinical Trial to Evaluate the Effectiveness of Abacavir 600 mg+ Lamivudine 300 mg as QD+ Efavirenz 600 mg QD Versus Kaletra 400/100 mg BID as Initial Antiretroviral Treatment
Brief Title: Study to Evaluate the Effectiveness of ABC+3TC +EFV in Once-Daily Regimens Versus KLT in Twice-Daily Regimens in Naive HIV Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Lluita Sida Foundation, Lluita Sida Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAKE; 2004-001282-18
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: HIV Infections
Keywords: Simplification therapy; Efficacy; Safety; Virological effectiveness; Immunological effectiveness; HIV
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Abacavir 600mg + lamivudine 300mg in on table QD + efavirenz 600mg QD
  Interventions: Drug: Kivexa
- B (Experimental): Abacavir 600mg + lamivudine 300mg in ine tablet QD * lopinavir/ritonavir 400/100 mg BID
  Interventions: Drug: Kivexa

INTERVENTIONS:
Drug: Kivexa — abacavir 600mg + lamivudine 300mg in one tablet QD

SUMMARY:
To evaluate the therapeutic equivalence between the two arms of treatment in virological and immunological response after 48 weeks and to evaluate the presence of side effects during the follow-up period.

DETAILED DESCRIPTION:
The efficacy of the highly active antiretroviral treatment (HAART) has been demonstrated in several clinical trials. Even so, a substantial proportion of patients do not manage to maintain correct viral suppression in daily clinical practice.

Adherence to HAART treatment is critical to obtain lasting viral suppression. Thus, factors that are related to adherence such as high pill load or takes, the complexity of the antiretroviral system, tolerability and food restrictions may have an effect on viral replication.

It has been demonstrated that simpler regimens with a scant number of tablets, without food restrictions and with a single take a day are safe, efficacious and that adherence improves.

The combination of abacavir 600 mg + lamivudine 300 mg QD in a single tablet is a novel dosage that may help increase treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years.
2. HIV-1 infected patients.
3. Naive to antiretroviral treatment.
4. Candidate patient for initiating antiretroviral treatment*.
5. Subject able to follow the treatment period.
6. Signature of the informed consent.
7. Women may not be fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use two contraceptive methods during the study, one of them at least being a barrier method.

Exclusion Criteria:

1. Hepatic tests > 5 times above normality.
2. Pregnancy or breastfeeding.
3. Treatment for opportunistic infections or neoplasms associated with the stable HIV over the last 6 weeks.
4. Suspected or documented resistance to any of the investigational drugs.
5. Known allergic hypersensitivity to any of the investigational drugs or any similar drug.
6. Subjects with abusive consumption of alcohol or illegal drugs.
7. Patients participating in another clinical trial.
8. Terminal renal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the virological response over the 48 weeks of the study. | At 12, 24, 36 and 48 weeks

SECONDARY OUTCOMES:
To evaluate the immunological efficacy (changes in CD4 and CD8 counts) of the combination studied over the follow-up period. | At 12, 24, 36 and 48 weeks.
To evaluate the impact of treatment on the lipid profile. | At 12, 24, 36 and 48 weeks
To evaluate the tolerance and safety of the combination of Efavirenz + lamivudine + abacavir given once daily over the 48-week treatment period. | At 12, 24, 36 and 48 weeks.
To evaluate treatment adherence (assessed by a self-reported questionnaire and with graduated satisfaction scales) and patient quality of life (assessed by means of the MOS-HIV questionnaire). | At 12, 24, 36 and 48 weeks.
To analyse the mutations that appear in patients that present virological failure. | When there is a virological failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit
Locations (20):
- Institute of Infections and Tropical Diseases University of Brescia, Brescia, Italy
- Spain (19):
  - Hospital Arquitecto Marcide, Ferrol, A Coruña
  - Hospital Generall de Alicante, Alicante, Alacant
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hopsital Gregorio Marañón, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hopsital Costa del Sol, Marbella, Malaga
  - Hospital Nuestra Sra del Rosell, Cartagena, Murcia
  - Hospital General de Murcia, Murcia, Murcia
  - Hospital Central de Asturias, Asturias, Oviedo
  - Hospital Xeral de Vigo, Vigo, Pontevedra
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital de Tarragona, Tarragona, Tarragona
  - Hospital Universitari Dr. Peset, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza